CLINICAL TRIAL: NCT02800655
Title: A Prospective Single Arm Open Label Intervention Study Using the DHFS With HIV Infected Participants Initiating or Continuing HIV Treatment
Brief Title: Digital Health Feedback System for Longitudinal Measurement of Medication Adherence During Anti-Retroviral (ARV)Therapy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of California, San Diego (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Gilead Sciences (Industry); ViiV Healthcare (Industry); GlaxoSmithKline (Industry); Proteus Digital Health, Inc. (Industry)
Responsible Party: Principal Investigator, Sara H. Browne, MD, MPH, Staff Research Associate, University of California, San Diego
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 160521; R01MH110057 (NIH)
Record Dates: First submitted 2016-04-05; First posted 2016-06-15 (Estimated); Last update posted 2022-12-23 (Actual); Status verified 2022-12

CONDITIONS: HIV
Keywords: ARV treatment; Medication Adherence; Digital Health Feedback System; Proteus Digital Health
MeSH Terms: conditions — Medication Adherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- DHFS with IS-ARV (Experimental): Digital Health Feedback System (DHFS) with either IS- Odefsey®, IS- Genvoya®, IS-Biktarvy®, IS- Tivicay® and Truvada® or IS- Tivicay® and Descovy ® (IS-co-encapsulated with ingestion sensor) -1 or 2 capsules daily (QD), depending on the treatment regimen, administered orally for 16 weeks.
  Interventions: Device: Digital Health Feedback System

INTERVENTIONS:
Device: Digital Health Feedback System — This intervention uses an ingestion sensor and a wearable sensor (worn as a patch on the skin), which are new technologies approved by the FDA, to collect information about patients taking their ARV medications. The wearable sensor records information, which is uploaded wirelessly to a mobile device and then to a secure computer. Together the sensors and the mobile device transmitting the information to the study computer are called a digital health feedback system (DHFS), which provides information about when patients have taken their ARV medications.
  Other Names:
  DHFS

SUMMARY:
This study uses an ingestion sensor and a wearable sensor (worn as a patch on the skin), which are new Proteus Digital Health (PDH) technologies approved by the FDA, to collect information about patients taking their ARV medications. The wearable sensor records information, which is uploaded wirelessly to a mobile device and then to a secure computer. Together the sensors and the mobile device transmitting the information to the study computer are called a digital health feedback system (DHFS), which gives healthcare providers information about when patients have taken their ARV medications.

The purpose of the study is to demonstrate that the DHFS is easy to use and acceptable to the HIV patient population; that patients will persist with its use; and that the system provides valid, accurate measures of adherence.

DETAILED DESCRIPTION:
This study is a prospective single arm open label intervention study over 16 weeks using the DHFS with ARV-naive subjects initiating HIV treatment. The study intervention has an initiation (Phase 1), persistence (Phase 2) and follow-up period up to 96 weeks. In phase 1 Subjects will use the DHFS with close follow-up incorporating visits with directly observed ingestions. In Phase 2 the Subjects utilize the DHFS in their natural setting with sporadic study visits until 16 weeks. Eligible HIV seropositive subjects who are at least 18 years of age, are HIV treatment naïve, and are initiating antiretroviral therapy prescribed by their HIV practitioner will receive an ingestible sensor enabled oral Anti-Retroviral or IS-ARV either IS-R/F/TAF (Odefsey®), IS-EC/F/TAF (Genvoya®), IS-BIC/F/TAF (Biktarvy®), IS-DTG/TDF/FTC (Tivicay® and Truvada®) or IS-DTG/TAF/FTC (Tivicay® and Descovy ®). The study will be conducted at the UCSD AVRC. Subjects will be recruited from UCSD AVRC, UCSD Owen Clinic, related or affiliated UCSD HIV primary care programs or community HIV primary care clinics. Following the 16 week intervention HIV plasma viral load and continuation in HIV care are followed for up to 96 weeks. The primary outcome will be an accurate measure of adherence i.e. the number of doses of selected IS-ARVs ingested, as captured by the DHFS, over the number of doses prescribed, adjusted for PDA. The investigators will also assess the acceptability and feasibility of longitudinal monitoring in real time of the ingestion rate utilizing the DHFS. In addition the investigators will evaluate the ability of the DHFS to identify subjects whose longitudinal medication taking and timing patterns in the first 16 weeks of ARV treatment puts them at risk for detectable HIV RNA levels as far out as 96 weeks from start of treatment.

PHARMACOKINETIC (PK) SUBSTUDY

A subset of 15 participants prescribed an IS-Dolutegravir regimen will be enrolled in a PK sub-study to generate a projected time-course of drug concentrations across the entire study period. On Day 14 of treatment sub-study participants will have a detailed PK profile for Dolutegravir obtained over a single dosing interval.

Participants will also have random plasma Dolutegravir levels measured at 4, 8, 12, and 16 weeks during the DHFS monitoring.Plasma HIV-1 RNA and CD4+ T-cell count will be measured at study entry.

At the start of the IS-Tivicay, participants included in the PK study will undergo intensive monitoring of viral decay dynamics with plasma HIV-1 RNA measured at baseline and Days 2, 7, 10 and 14, as well as at Weeks 4, 8, 12, and 16 to provide the dynamic range of virologic suppression relative to drug exposure profiles generated from the intensive PK sampling on Day 14 and the DHFS dosing history.

ELIGIBILITY:
Inclusion Criteria:

1. HIV seropositive status, as documented by positive licensed HIV antibody testing AND either treatment naïve, defined as never having received ARVs in the past (excluding ARVs used as pre-exposure prophylaxis OR post-exposure prophylaxis) or continuing HIV treatment.
2. Persons ready to initiate first regimen treatment for HIV infection by their HIV provider, that includes either:

   * Biktarvy®
   * Genvoya®
   * Odefsey®
   * Tivicay® PLUS Truvada®
   * Tivicay®: PLUS Descovy®
3. Eligible for antiretroviral medications and in possession of prescriptions for above noted study eligible regimens.
4. Laboratory values obtained by screening laboratories within 30 days of entry:

   * Absolute neutrophil count (ANC) ≥ 1,000/mm3.
   * Hemoglobin ≥ 9.0 g/dL.
   * Platelet count ≥ 75,000/mm3.
   * AST (SGOT), ALT (SGPT), and alkaline phosphatase ≤ 3 x ULN.
   * Total bilirubin ≤ 1.5 x ULN and direct bilirubin.
   * Estimated GFR by Cockcroft-Gault equation of greater than 50 ml/min, if starting treatment with Tivicay®: Dolutegravir (DTG) PLUS Truvada®: Tenofovir disoproxil fumarate/Emtiritabine (TDF/FTC)
   * Estimated GFR by Cockcroft-Gault equation of greater than 30 ml/min, if starting treatment with Genvoya®: Elvitegravir/Cobisistat/Tenofovir alafenamide/Emtricitabine (E/C/F/TAF), Biktarvy®(BIC/F/TAF), Odefsey®: Riplivirine/Tenofovir alafenamide/Emtricitabine (R/F/TAF), or with Tivicay®: Dolutegravir (DTG) PLUS Descovy®: Tenofovir alafenamide/Emtricitabine (F/TAF)
   * HIV RNA value (viral load) ≤ 100,000 copies/mL, if starting treatment with Odefsey®: Riplivirine/Tenofovir alafenamide/Emtricitabine (R/F/TAF)
5. Females of childbearing potential must agree to use an acceptable form of contraception throughout the protocol and for 6 weeks after stopping the IS-ARV medications.
6. Men and women age ≥ 18 years.
7. Basic competency in understanding written and verbal information as it applies to DHFS use. English and Spanish will be used for study documents and communication.
8. Willing to follow all protocol requirements.
9. Ability to use mobile device per investigator determination, and to wear PDH wearable sensor (i.e., no skin conditions precluding use).
10. Ability and willingness of subject to give written informed consent.

    -

Exclusion Criteria:

1. Female who is pregnant, breast-feeding, or of childbearing potential and disagrees to use contraception throughout the study period.
2. Use of any of the prohibited medications or other non-informed medications (Section 5.5.2) within 30 days of study entry (Day 0).
3. Known allergy/sensitivity to any of the study drugs.
4. Known sensitivity to skin adhesives.
5. Serious medical (serious infection or acute therapy for other medical illness) or psychiatric illness requiring systemic treatment and/or hospitalization until subject either completes therapy or is clinically stable on therapy, in the opinion of the investigators, for at least 30 days prior to study entry (Day 0).
6. Evidence of any major antiretroviral resistance associated mutation in genotypic testing at baseline, prior to study entry for subjects. Resistance testing results must be available for review by the site investigator and study protocol team prior to enrollment to ensure that no exclusionary resistance exists. All resistance testing results should be scanned and uploaded to the on-line data collecting system (https://cfar.ucsd.edu/intranet).

   NOTE: Subjects will be excluded if genotype shows presence of any HIV-associated resistance mutations listed per the International AIDS Society-USA mutation list (update lists can be found at: http://www.iasusa.org).
7. Active drug or alcohol use, or dependence, or other conditions that, in the opinion of the site investigators, would significantly interfere with ability to follow to study requirements.
8. History of pancreatitis

   -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-06; Primary Completion 2021-12 (Actual); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Medication taking adherence | 16 weeks
  Medication taking adherence, defined as the number of doses ingested as captured by the DHFS over the number of doses prescribed, adjusted for Positive Detection Accuracy ( determined by the percentage of HIV medication ingestion detected by the DHFS administered under witnessed observation).

SECONDARY OUTCOMES:
The persistence of sensor-enabled ingestions | 16 weeks
  Defined as the number of detected ingestion divided by the number of expected ingestions, over the duration of monitoring.
Participants will be classified into groups according to the accurate measurement of adherence | 16 weeks
  High 95-100% adherence, Normal 90-95% adherence, At risk 80-90% taking adherence, Severe Risk <80%
Medication behavior during IS-ARV use | 16 weeks
  Defined as the overall number of doses taken divided by the number of expected doses and by patterns of medication behavior (timing of dose, patterns of skipped doses, doses related to physiological parameters).

CONTACTS AND LOCATIONS:
Overall Officials: Sara H Browne, MD, MPH, Study Chair — University of California, San Diego AntiViral Research Center; Constance A Benson, MD, Study Chair — University of California, San Diego AntiViral Research Center
Locations (2):
- United States (2):
  - Family Health Centers of San Diego, San Diego, California
  - UCSD AntiViral Research Center, San Diego, California

IPD SHARING:
Plan to Share IPD: Yes